CLINICAL TRIAL: NCT00003769
Title: A Phase II Trial of Perillyl Alcohol in Patients With Resectable Pancreatic Cancer
Brief Title: Perillyl Alcohol Followed by Surgery in Treating Patients With Stage II or Stage III Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Patrick Loehrer, MD/ Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Purpose: Treatment
Other Study IDs: 9710-07; T98-0046; IUMC-9710-07; NCI-T98-0046
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — perillyl alcohol; Surgical Procedures, Operative

INTERVENTIONS:
Drug: perillyl alcohol
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of perillyl alcohol followed by surgery in treating patients who have stage II or stage III pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the biologic activity of perillyl alcohol in patients with potentially resectable, stage II or stage III pancreatic adenocarcinoma. II. Characterize the acute toxicity of this drug in these patients. III. Evaluate the antitumor activity of this drug in these patients. IV. Monitor and quantitate the plasma levels of perillyl alcohol after oral administration in this patient population.

OUTLINE: Patients receive oral perillyl alcohol 4 times daily on days 1-14. Patients undergo surgical resection on day 15. There is no continuation of perillyl alcohol postoperatively. Patients are followed at a minimum of 2 and 4 months following surgery.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage II or stage III pancreatic adenocarcinoma that is considered resectable Lesions should be amenable to surgery with curative intent Bidimensionally measurable or evaluable disease No evidence of metastatic disease No clinically detectable third space fluid collections (e.g., ascites or effusions)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.5 g/dL Hepatic: Bilirubin no greater than 4 times upper limit of normal (ULN) PTT no greater than 1.5 times control (unless on anticoagulants) Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception No concurrent serious systemic disorders incompatible with study No active infection No second primary malignancy, previously untreated with curative intent or presently active, that would preclude curative resection of the pancreas

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for pancreatic carcinoma Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for pancreatic carcinoma Surgery: See Disease Characteristics Other: At least 1 month since prior investigational agents At least 72 hours since prior anticoagulant therapy, cholesterol-lowering agents (e.g., lovastatin), high dosage vitamins, or antioxidants No concurrent anticoagulants except for the sole purpose of central line patency maintenance No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Loehrer, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States